CLINICAL TRIAL: NCT03011684
Title: Fertility Preservation Using Tamoxifen and Letrozole in Estrogen Sensitive Tumors Trial
Acronym: TALES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TALES Trial; NCI-2017-01809 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 16751 (Other: University of California, San Francisco)
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Infertility
Keywords: Fertility Preservation; Breast Cancer
MeSH Terms: conditions — Infertility; Breast Neoplasms | interventions — Tamoxifen; Letrozole

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at the time of enrollment to 1 of 2 experimental arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Randomized ER Positive Participants (Letrozole) (Experimental): Participants will receive 5 mg of letrozole with the first day of non-investigational gonadotropin (letrozole-gonadotropin) and stopped on the day of oocyte retrieval.
  Interventions: Drug: Letrozole
- Randomized ER Positive Participants (Tamoxifen) (Experimental): Participants will receive 20 mg of tamoxifen with the first day of non-investigational gonadotropin (tamoxifen-gonadotropin) and stopped on the day of oocyte retrieval
  Interventions: Drug: Tamoxifen
- ER Negative (ER-) Participants (No Intervention): Participants whose disease is ER negative will be consented and used as a reference cohort and will receive no study related medication. The Gonadotropin received is non-investigational and part of usual care.

INTERVENTIONS:
Drug: Tamoxifen — Given orally
  Other Names: Nolvadex; Soltamox
  Arms: Randomized ER Positive Participants (Tamoxifen)
Drug: Letrozole — Given orally
  Other Names: Femara
  Arms: Randomized ER Positive Participants (Letrozole)

SUMMARY:
Latrogenic infertility as a result of cancer treatment has a profound effect on long-term quality of life in survivors of reproductive-age cancers. Oocyte cryopreservation prior to cancer treatment has been associated with improved quality of life, with a potential ability to reduce long-term decision-related regret in cancer survivors. Though letrozole plus gonadotropin and and tamoxifen plus gonadotropin are currently routinely used worldwide in ovarian stimulation cycles for fertility preservation in patients with estrogen-receptor-positive breast cancer, it is not clear which of the two might lead to improved oocyte yield. Improved knowledge about the efficacy of these medications, with regard to oocyte yield, has the potential to significantly improve quality of life in reproductive-age breast cancer survivors.

DETAILED DESCRIPTION:
Purpose:

Our primary objective is to determine whether concomitant administration of tamoxifen 20 mg oral with gonadotropins (tamoxifen-gonadotropin) versus a starting dose of letrozole 5 mg oral with gonadotropins (letrozole-gonadotropin) will result in a difference in mature oocyte yield during our routine ovarian stimulation protocol for fertility preservation for Estrogen-Receptor-Positive (ER+) breast cancer.

Specific Aims: Each of the following aims will include a primary comparison and secondary comparisons.

Primary aim: The primary aim will be to compare patients with ER+ breast cancer who are treated with letrozole-gonadotropin versus patients with ER+ breast cancer who are treated tamoxifen-gonadotropin with regard to ovarian stimulation outcomes.

* Primary comparison:

  1) To determine if the assigned stimulation regimen will result in a difference in mature (meiosis II) oocyte yield in patients with breast cancer who undergo ovarian stimulation for fertility preservation.
* Secondary comparison:

  1. To compare estrogen, progesterone, and androgen levels during the ovarian stimulation cycle.
  2. To compare estrogen, letrozole, and tamoxifen levels in follicular fluid.
  3. To compare duration of stimulation (days) and total gonadotropin dose (international units of FSH).
  4. To assess embryo quality, if applicable, on day 3 and day 5 of embryo culture, a measure of the developmental competence of the oocytes.
* Experimental comparison:

  1. To compare clinical pregnancy rates when cryopreserved tissue is eventually utilized among patients from the assigned stimulation regimens. This comparison is labeled experimental because of the remoteness of such an outcome from our present study.

Secondary Aim: We will repeat the above comparisons among patients with ER+ breast cancer who are treated with tamoxifen-gonadotropin versus a prospectively-obtained reference group of patients with Estrogen-Receptor-Negative (ER-) breast cancer who are treated gonadotropin alone. We will then again repeat the above comparisons among patients with ER+ breast cancer who are treated letrozole-gonadotropin versus patients with ER- breast cancer who are treated gonadotropin alone.

Experimental Design and Methods:

Study population:

The target population is reproductive-age women who have been recently diagnosed with ER+ breast cancer and choose to undergo oocyte or embryo cryopreservation prior to chemotherapy treatment. All eligible women will be asked to join the study at their initial University of California, San Francisco (UCSF) fertility preservation consult. Study participants will be recruited from the Reproductive Endocrinology Clinic at University of California, San Francisco Center for Reproductive Health. A consecutive sample with ER- disease will also be recruited at the same type of visit. They will be asked to take part in the gonadotropin only stimulation group, which will be used for a secondary aim.

ELIGIBILITY:
Inclusion Criteria:

* New breast cancer diagnosis
* Has not yet begun chemotherapy
* Desires to undergo ovarian stimulation and oocyte retrieval prior to cancer treatment
* Age 18 years old or greater

Exclusion Criteria:

* Chemotherapy has already commenced or been completed
* History of recurrent breast cancer (with a prior history of chemotherapy)
* Stage IV breast cancer diagnosis (metastases remote from the breast)
* Patient's oncologist advises against the trial - in which case they can choose to receive stimulation with letrozole+gonadotropin
* Does not plan to undergo ovarian stimulation and oocyte retrieval prior to diagnosis
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up, or interpretation of study results
* Age less than 18 years old

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 309 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mature Oocyte Yield | Up to 2 weeks
  To determine if the assigned stimulation regimen will result in a difference in mature (meiosis II) oocyte yield in patients with breast cancer who undergo ovarian stimulation for fertility preservation. An Effect Size of 3 mature oocytes, based on clinically significant difference of 2 embryos to transfer. An average of 2 embryos are transferred per freeze-thaw cycle. If ~75% of mature oocytes will become embryos that can be frozen, then 3 mature oocytes should yield ~2 embryos for transfer. This effect size would effectively mean an additional event of embryos transferred.

SECONDARY OUTCOMES:
Compare change in estrogen levels during the ovarian stimulation cycle | Up to 2 weeks
  Estrogen level data will be collected at baseline and after completion of the stimulation cycle
Compare change in progesterone levels during the ovarian stimulation cycle | Up to 2 weeks
  Progesterone level data will be collected at baseline and after completion of the stimulation cycle
Compare change in androgen levels during the ovarian stimulation cycle | Up to 2 weeks
  Androgen level data will be collected at baseline and after completion of the stimulation cycle
Compare change in estrogen in follicular fluid | Up to 2 weeks
  Estrogen levels in follicular fluid will be collected at baseline and after completion of the stimulation cycle
Compare change in letrozole in follicular fluid | Up to 2 weeks
  Letrozole levels in follicular fluid will be collected at baseline and after completion of the stimulation cycle
Compare change in tamoxifen in follicular fluid | Up to 2 weeks
  Tamoxifen levels in follicular fluid will be collected at baseline and after completion of the stimulation cycle
Compare duration of stimulation (days) and total gonadotropin dose | Up to 2 weeks
  The duration of stimulation in days will be compared to total gonadotropin dose across all groups.
Number if competent oocytes on day 3 of embryo culture | Up to 2 weeks
  To assess embryo quality, if applicable, on day 3 of embryo culture, a measure of the developmental competence of the oocytes.
Number if competent oocytes on day 5 of embryo culture | Up to 2 weeks
  To assess embryo quality, if applicable, on day 5 of embryo culture, a measure of the developmental competence of the oocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California at San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Letourneau J, Juarez-Hernandez F, Wald K, Ribeiro S, Wang A, McCulloch CE, Mok-Lin E, Dolezal M, Chien AJ, Cedars MI, Rosen M. Concomitant tamoxifen or letrozole for optimal oocyte yield during fertility preservation for breast cancer: the TAmoxifen or Letrozole in Estrogen Sensitive tumors (TALES) randomized clinical trial. J Assist Reprod Genet. 2021 Sep;38(9):2455-2463. doi: 10.1007/s10815-021-02273-3. Epub 2021 Jul 26. PMID 34312774